CLINICAL TRIAL: NCT05231967
Title: The Predictive Value of the Left Atrial Kinetic Energy for Atrial Fibrillation Recurrence
Brief Title: Bursa Postgraduate Hospital Department of Cardiology
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Professor Doctor, Bursa Postgraduate Hospital
Other Study IDs: Bursa Postgraduate Hospital AF
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial fibrillation recurrence: Atrial fibrillation recurrence one month after cardioversion
  Interventions: Other: Cardioversion
- Sinus rhythm continue: Sinus rhythm continue one month after cardioversion
  Interventions: Other: Cardioversion

INTERVENTIONS:
Other: Cardioversion — In proper atrial fibrillation patients, cardioversion was performed to provide sinus rhythm

SUMMARY:
Ensuring and maintaining normal sinus rhythm is critical for reducing negative outcomes in patients with atrial fibrillation (AF). Electrical direct current cardioversion is a frequently used method of restoring SR, but a significant proportion of patients later develop AF recurrence. Determining which of these patients is prone to recurrence is important for treatment modification. Left atrial kinetic energy (LAKE) is a parameter that shows left atrial mechanical function and can be calculated noninvasively by transthoracic echocardiography. LAKE is reduced in patients with AF recurrence.

DETAILED DESCRIPTION:
Study population: The study was initiated after the ethics committee of Bursa Postgraduate Hospital approved the study protocol. A total of 120 consecutive patients aged 18 years and older who underwent successful electrical cardioversion following persistent atrial fibrillation (AF) were included in the study. Persistent AF was defined as continuous AF lasting longer than seven days in electrocardiography follow-up (9). Patients with significant valvular disease, previous valve surgery, severe left ventricular systolic dysfunction (ejection fraction < 40%), severely dilated left atrium (> 5 cm), previous ablation of atrial fibrillation, or paroxysmal atrial fibrillation were excluded from the study.

The patients were divided into two groups - patients who remained in sinus rhythm (SR) (group 1) and patients with AF recurrence (group 2) after one month of follow-up.

Echocardiography: All patients underwent routine transthoracic echocardiography (TTE) prior to cardioversion and transoesophageal echocardiography (TEE) (EPIQ 7 Echocardiography Machine, Philips Ultrasound, Netherlands) to exclude left atrial and left atrial appendage thrombus. TTE was repeated in patients who remained in SR 24 hours after cardioversion. All standard measurements were taken from the parasternal long and short axes and apical two- and four-chamber windows. All assessments and measurements were made according to the American Society of Echocardiography (ASE) guidelines (10).

Left ventricular ejection fraction (LVEF) was calculated according to the modified biplane Simpson method (10). Mitral flow velocities were recorded from the apical four-chamber view with a sample volume of 5 mm placed at the level of the mitral valve tips using pulsed-wave Doppler (PWD). Peak early (E) and late (A) mitral entry velocities were recorded.

LAKE (left atrial kinetic energy) values were calculated at the 24th hour after cardioversion. LAKE was defined as 0.5 × left atrium stroke volume (cm³, volume at the beginning of left atrial systole - left atrium minimal volume) × 1.06 (g/cm³, blood density) × (peak A velocity)² (cm/sec, transmitral PWD A velocity) (8).

ELIGIBILITY:
Inclusion Criteria:

* persistent atrial fibrillation
* underwent successful electrical cardioversion
* suitable for echocardiographic imaging
* who agreed to participate in the study

Exclusion Criteria:

* significant valvular disease,
* previous valve surgery,
* severe left ventricular systolic dysfunction (ejection fraction < 40%),
* severely dilated left atrium (> 5 cm),
* previous ablation of atrial fibrillation, or paroxysmal atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persistent atrial fibrillation patients.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
sinus rhythm continue one month after cardioversion | one month
  atrial fibrillation recurrence

IPD SHARING:
Plan to Share IPD: Undecided